CLINICAL TRIAL: NCT03342079
Title: Effectiveness of Nitrous Oxide 50% for Reducing Pain and Distress Associated with Needle-stick in Children: a Prospective Randomized Blinded Controlled Trial
Brief Title: Effectiveness of Nitrous Oxide 50% for Reducing Pain and Distress Associated with Needle-stick in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Boston Children's Hospital (Other)
Collaborators: Linde AG (Industry)
Responsible Party: Principal Investigator, Navil Sethna, Anesthesiologist, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P00002478
Record Dates: First submitted 2017-06-12; First posted 2017-11-14 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2023-11

CONDITIONS: Local Anesthetic Efficacy
MeSH Terms: interventions — Tetracaine; Transdermal Patch; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (3):
- Group 1 (Experimental): local anesthetic (lidocaine 70 mg/tetracaine 70 mg topical patch; Synera) + placebo
  Interventions: Drug: Local Anesthetics,(lidocaine 70 mg/tetracaine 70 mg topical patch; Synera); Drug: Placebos
- Group 2 (Experimental): local anesthetic (lidocaine 70 mg/tetracaine 70 mg topical patch; Synera) + nitrous oxide
  Interventions: Drug: Local Anesthetics,(lidocaine 70 mg/tetracaine 70 mg topical patch; Synera)
- Group 3 (Placebo Comparator): Placebo + nitrous oxide
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Local Anesthetics,(lidocaine 70 mg/tetracaine 70 mg topical patch; Synera) — topical anesthetic (lidocaine 70 mg/tetracaine 70 mg topical patch; Synera)
  Other Names: Synera
  Arms: Group 1; Group 2
Drug: Placebos — placebo topical anesthetic
  Other Names: Synera patch without local anesthetics
  Arms: Group 1; Group 3

SUMMARY:
Venipuncture (puncturing of a vein) through the skin in order to insert a vein catheter (also know as cannula) is one of the most common needle-related medical procedures performed in children. Venipuncture is necessary for administration of sedation to facilitate motionless patient state for radiological imaging studies such as diagnostic nuclear medicine imaging or CT scan studies.

The current practice for management of needle-related pain is to use needle-less topical local anesthetic delivery systems. These delivery systems are increasingly used in children to anesthetize the skin prior to venipuncture and venous cannulae insertion. This can reduce the pain and distress associated with the needle sticks, however, many children express considerable fear, anxiety and distress during medical procedures that involve needles. Anticipatory pain and phobia associated with needle stick may render the patient uncooperative and anxious even when effective analgesia is produced by a topical local anesthetic.

Both the discomfort and associated anxiety during such an intervention can be considerably improved when inhaled nitrous oxide is used alone or in combination with local anesthetics. The administration of nitrous oxide (50% to 70%) for painful procedures is an effective and safe method of suppressing procedural pain and distress in children over the age of one year (level 3 evidence). When compared to other intravenous sedation agents, nitrous oxide 50% used for uncomplicated painful procedures is associated with markedly shorter recovery time and less respiratory side effects (level 3 evidence). When combined with local anesthetics for procedural pain and stress management, nitrous oxide 50% is more effective and has higher success rate compared to orally administered anxiolytics or local anesthetic alone (level 2 evidence). Combining nitrous oxide (50-70%) and local anesthetics is shown to be a more effective procedural sedation than local anesthetics alone (level 1 evidence).

The efficacy and safety of inhaled 50-70% nitrous oxide for relief of mild-to-moderate anxiety and pain of venipuncture in children just prior to induction of anesthesia have been investigated in randomized controlled trials by anesthesiologists; physician who are skilled and competent in providing optimal sedation in the operating room setting. The major benefit of administration of a fixed low concentration of 50% nitrous oxide for procedural sedation is that it achieves pain relief while retaining verbal contact with the patient. The efficacy, safety and tolerability of administration of low fixed concentration 50% nitrous oxide using a nitrous oxide mask delivery system for control of mild-to-moderate procedural sedation during performance of needle-related pain (i.e., venipuncture) in children has not been investigated in a blinded randomized controlled trials outside the operating room setting when provided by skilled and competent non-anesthesia trained personnel.

In view of safety of low concentration (50%) of nitrous oxide due to preservation of the patent airway, lack of respiratory depression and rapid recovery, investigators propose this preliminary study to validate the hypothesis that nurse-administered premixed inhaled nitrous oxide and oxygen at a fixed 50:50% concentration with or without a topical anesthetic can provide safe and effective pain relief and reduce behavioral distress in preschool children during routine placement of intravenous cannulation prior to administration of intravenous sedation for nuclear medicine studies and CT imaging studies.

To test this hypothesis, investigators propose performing a prospective, double blind control trial in 105 children undergoing nuclear medicine studies or CT imaging, randomized into three groups;

1. the treatment groups will receive either nitrous oxide and a placebo topical anesthetic patch or
2. nitrous oxide and a topical anesthetic patch (Synera) and
3. the placebo group will receive oxygen mask and a topical anesthetic patch (Synera).

The topical anesthetic patch or placebo patch will be applied for 20 minutes prior to the scheduled insertion of intravenous cannula. The use of a topical local anesthetic such as the Synera patch is a standard of care for placement of intravenous cannula at Children's Hospital Boston.

Assessments to estimate the effectiveness of nitrous oxide with and without the use of topical anesthesia Synera patch will include;

1. Assessment of child's pain and observer report of pain control.
2. Child's anxiety before and during the procedure.
3. Tolerability of the mask delivery system of a fixed concentration of 50% nitrous oxide outside the operating room.
4. Accuracy of nitrous oxide delivery dose by measuring the end-tidal concentration of nitrous oxide.
5. Adverse events related to use of nitrous oxide alone or in combination with a topical analgesic.

DETAILED DESCRIPTION:
This study was never conducted due to lack of funding

ELIGIBILITY:
Inclusion Criteria:

* • Children ages 3 to 6 years of age who require diagnostic CT or nuclear medicine studies under conscious sedation

  * Guardians give consent and the child gives assent when appropriate
  * Both genders
  * All racial and ethnic groups
  * English and other languages speaking and reading children and guardians (for consent/assent purposes)

Exclusion Criteria:

* Age less than 3 or older than 6 years

  * Patients who had a history of adverse events with facemask; mask phobia
  * If parents/patients refuse to participate in the study
  * Fasting less than 2h for clear liquids, 4h breast milk, 6h formula and fortified breast milk for under 1 yr and 8h for over 1yr, 8h for non-human milk and solid food.
  * Impairment of cognition/neurologic, hepatic, renal, cardiovascular, endocrine, metabolic, and/or coagulation function.
  * A history of any diagnosis of psychiatric disorders as reported by parents/guardians
  * A history of chronic pain and/or use of chronic (daily around the clock) opioids, other analgesics or sedatives/hypnotics
  * Intake of prescription medications or over-the-counter medications known to affect pain perception such as narcotics, non-steroidal anti-inflammatory agents, stimulants, hypnotics, sedatives, etc. within 8 hours of planned surgical procedure
  * Vitamin B12 & folate deficiency
  * Immune suppression (e.g., postoperative organ transplant, chemotherapy, neutropenia, any condition suppresses immunity or bone marrow)
  * Abnormal homocysteine metabolism
  * Lung cyst, bowel obstruction, middle ear disease, pneumothorax, head injury, active gastro-esophageal reflux, history of delayed gastric emptying and vomiting, upper airway obstruction, airway infection, active wheezing from asthma, and apnea
  * Significant impairments: pulmonary hypertensions, cardiomyopathy, hypovolemia, meningitis, space occupying lesions of the brain e.g. tumors, sepsis, severe liver diseases (e.g., biliary atresia, liver failure)

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Analgesia measured using the Observational Visual Analog Pain Assessment Scale (0= no pain and 10= unimaginable severe pain) | During venipuncture procedure
  decrease pain during venous blood drawing

IPD SHARING:
Plan to Share IPD: No